CLINICAL TRIAL: NCT00343499
Title: A Single Center, Randomized Trial to Evaluate the Effects of Diovan to Maintain Sinus Rhythm in Patients With Persistent Atrial Fibrillation
Brief Title: The Use of DIOVAN to Reduce Post-Cardioversion Recurrence of Atrial Fibrillation Trial (the DRAFT Trial)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inability to recruit
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 128-011
Record Dates: First submitted 2006-06-21; First posted 2006-06-23 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2008-08

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; valsartan; sinus rhythm; persistent atrial fibrillation undergoing electrical cardioversion to restore normal sinus rhythm
MeSH Terms: conditions — Atrial Fibrillation | interventions — Valsartan

INTERVENTIONS:
Drug: valsartan

SUMMARY:
24 week, single center, prospective, randomized, double-blind treatment study of valsartan (80 mg/bid, increased to 160 mg/bid) or placebo in addition to other general medical therapy in patients with persistent atrial fibrillation (AF) undergoing electrical cardioversion to restore normal sinus rhythm (SR).

DETAILED DESCRIPTION:
To evaluate the efficacy of valsartan, added to standard AF therapy, to maintain sinus rhythm and extend the interval to first AF recurrence after cardioversion.Evaluate the efficacy of valsartan, begun prior to cardioversion, on the difficulty (number and total energy of CV attempts), the net rate of cardioversion (to SR for >10 minutes), and early AF recurrence rate (within 24 hours)

ELIGIBILITY:
Inclusion Criteria:

* The patient (male or non-pregnant female) must be >18 years of age
* Have ECG documented AF at the time of enrollment into the study
* Require (be scheduled for) electrical cardioversion
* Female patients of childbearing potential must have a documented negative pregnancy test during the index hospitalization.
* The patient or legally authorized representative willing to give written informed consent, prior to the procedure, using the ICF approved by the UCR Institutional Review Board. Surrogate consent must be given per CV Research SOP.
* Have a serum potassium level between 3.5 and 5.5 meq/L
* If diabetic, have a hemoglobin A1C level <11%
* NYHA I-II can be enrolled if no hospitalizations for heart failure within 6 months or current, known EF<40%.

Exclusion Criteria:

* The patient is unable or unwilling to cooperate with the study follow-up procedures.
* Pregnant and/or lactating women, and women of child bearing potential not using acceptable means of contraception. Women of childbearing potential must be using adequate measures of contraception (as determined by the Investigator) to avoid pregnancy and should be highly unlikely to conceive during the study period. Women of childbearing potential must have a negative pregnancy test at screen.
* Participation in any other clinical trials involving investigational or marketed products within 30 days prior to entry in the study.
* Current diagnosis of angina pectoris (no events within a period of 3 months prior to Visit 1 (V1)
* History or current diagnosis of symptomatic heart failure (NYHA classes III-IV) or
* documented ejection fraction of < 40 %. Myocardial Infarction within 3 months; coronary revascularization (PCI or CABG), unstable angina within 1 month of V1.
* Stroke, deep vein thrombosis (DVT), pulmonary embolism (PE) or transient ischemic attack (TIA) within 3 months of V1.
* Substance or alcohol abuse within 6 months of V1
* Known allergy to any of the drugs administered in the study (angiotensin receptor blocker (ARB) or an angiotensin converting enzyme inhibitor (ACE-I), Valsartan, amiodarone, flecainide or propafenone)
* Any other contraindication listed in the labeling of warfarin or acenocoumarol.
* Patients treated with ARBs or ACE-I within 1 month of V-1
* Impaired renal function defined as a serum creatinine > 2.5 mg/dL
* Evidence of hepatic disease evidenced by an AST or ALT value > 2 times the upper limit of the institution's normal values.
* Significant non-cardiovascular illness or condition likely to result in severe incapacitation or death prior to study completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2004-11; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Time to first AF recurrence on valsartan vs. placebo (time-to-event analysis, log-rank test)

SECONDARY OUTCOMES:
Number of CV attempts in order to restore SR in valsartan vs. placebo
Total electrical energy expended in 2 groups to achieve SR
Rate of early AF recurrence (within 24 hours) in the 2 groups after achieving SR
Net rate of NSR in the 2 groups at 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Anderson, MD, Principal Investigator — Intermountain Healthcare, LDS Hospital
Locations (3):
- United States (3):
  - McKay Dee Hospital, Ogden, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah